CLINICAL TRIAL: NCT04241848
Title: Use of a Powered Orthotic Exoskeleton to Promote Mobility Through Improved Squat, Knee Flexion and Loading of the Paretic Leg in Persons With Chronic Stroke
Brief Title: Powered Orthotic Exoskeleton Training in Stroke
Acronym: POETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3299-P; I21RX003299 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-27 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Exoskeleton Device; Walking; Neurological Rehabilitation; Paresis; Hemiplegia
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Ambulation training while using the powered orthotic exoskeleton for 36 sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Powered Orthotic Exoskeleton Training Group (Experimental): Participant in 36 session ambulation training using a powered orthotic exoskeleton.
  Interventions: Device: Keeogo; Other: Ambulation training
- Control Group (Active Comparator): Participant in 36 session ambulation training without using a powered orthotic exoskeleton.
  Interventions: Other: Ambulation training

INTERVENTIONS:
Device: Keeogo — A new and novel type of robotic-device (Keeogo, B-temia, Inc.) was developed to provide powered assistance at the knee for persons with stroke. This device provides assistance for both knee extension and knee flexion during ambulation, transfers to standing and sitting, in addition to ascending and descending stairs. As this device isn't able to fully control the movement, it requires the ability of the patient to stand and initiate stepping. The approach the Keeogo uses to monitor the desired movement in order to appropriately provide assistance. This promotes intuitive learning for the user, minimizing the amount of instruction and practice needed to effectively ambulate allowing users to independently ambulate within one session. This device does not restrict leg movement, so the user can side-step and walk backwards. However, it does not provide assistance during these movements.
  Arms: Powered Orthotic Exoskeleton Training Group
Other: Ambulation training — Ambulation training will consist of mobility activities affecting daily life including: walking; squatting (or getting in and out of a chair); bending, kneeling or stooping (for picking an item up off of the floor); and ascending and descending stairs. Sessions will be monitored and tailored to the individual, based on their functional ability and to ensure their safety.

SUMMARY:
Veterans who suffer strokes often have disturbances in the ability to walk that reduces independence and quality of life. Alterations in gait combined with general decreased activity are associated with reduced muscle strength of the paretic leg. This leads to cardiovascular deconditioning and reduced quality of life. There is a new and novel battery powered device (Keeogo powered orthotic exoskeleton) that uses motors that assist knee movement while walking, sitting down, and standing up. The Keeogo monitors hip movement to assist the knee, making it simple to learn how to use. If successful, this project will show how this device will help improve the ability to walk and provide evidence to support larger clinical trials in a home and community setting to improve mobility, increase muscle mass and strength in the legs, as well as improve general health and quality of life. Lastly, this device could be used to increase motivation and confidence in a person to walk for longer periods of time and distance, providing the ability to walk in places that were previously inaccessible.

DETAILED DESCRIPTION:
Ninety percent of stroke survivors have clinically significant gait impairments that lead to secondary medical complications, including cardiovascular deconditioning and reduced quality of life (QOL). Several rehabilitative interventions that increase the level of activity and mobility have been shown to be beneficial. Challenges posed by most of these locomotor gait training interventions require recurring visits to a rehabilitation center. The recent development of novel powered exoskeletons offers a potential mechanism for stroke survivors to improve mobility in the home and community. Although the predominant research using these devices have been in persons with spinal cord injury, there are currently two devices are commercially available for use in patients with stroke and additional devices are being developed. The Keeogo powered orthotic exoskeleton is a novel device intended for persons with stroke who can ambulate but have gait impairment. This device consists of a ridged orthotic structure placed over clothing on the legs and batteries to the power motors that assist both knees in gait movement. The system monitors hip movement driven by the user and interprets this movement to apply the appropriate assistance at the knee joint. This unique approach makes learning intuitive, enabling the user only to acclimate to the system rather than learning how to control the device to initiate the desired movement.

This proposal is a randomized controlled pilot study. Fifteen veterans with chronic stroke (>6months) and who retain some ability to take steps but have impaired gait will be recruited. Ten participants will be randomized into the exoskeleton group and 5 into the control group. Both groups will be asked to complete 36 one-hour sessions of ambulation training. The exoskeleton group will train using the Keeogo powered orthotic exoskeleton and the control group will train without using their own conventional aide.

The primary aim is to determine the efficacy of training with this exoskeleton and its ability to improve transfers to standing and sitting as assessed by the five times sit-to-stand test. A secondary aim will be to assess effects of the device during overground ambulation. Outcome measurements to investigate changes of knee range of motion and loading of the paretic limb. An exploratory outcome of changes in energy expenditure during ambulation with and without the powered exoskeleton. Additional exploratory outcome measures of QOL will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Males and female between 18 and 89 years old;
* Hemiplegia or hemiparesis due to stroke (>6 months);
* [Able to walk between 0.15-0.75m/s]
* Self-reported limitations to mobility and walking activities due to paretic side knee stiffness and loss of range of motion;
* Weight under 250lbs
* Desire to increase daily activity levels; and
* Able and willing to commit to participation and follow directions and communicate basic needs.

Exclusion Criteria:

* Neurological paralysis causing an inability to stand, weight bear or take stepping movements;
* Fixed contractures resulting in limited range of motion in the hip, knees, or ankles that prevent sitting, standing, walking, and/or squatting activities;
* Modified Ashworth Scale for spasticity greater than 3 in the lower limbs
* Able to walk at a normal walking speed (1.4 m/s, 3.2 mph) or better during the Six Minute Walk Test (6MWT)
* Anthropometric incompatibility with the device

  * Femur length less than 36 cm or greater than 45 cm;
  * Upper thigh circumference less than 55 cm or greater than 75 cm;
  * Lower thigh circumference less than 27 cm or greater than 40 cm;
  * Calf circumference less than 33 cm or greater than 49 cm;
  * Ankle circumference less than 27 cm or greater than 40 cm;
  * Shin length less than 26 cm;
  * Waist circumference less than 71 cm or greater than 107 cm;
* Any medical complication or co-morbidity as judged by the study physician to be contraindicated for wearing the device or walking (e.g., cardiovascular disorders, pressure ulcers, open wounds, lower limb vascular disorders, or other medical conditions); and
* Pregnant or planning to become pregnant (Females only).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Spungen, EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Where practicable, sharing should take place under a written agreement prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. However, it is permissible for final datasets in machine-readable format to be submitted to and accessed from PubMed Central (and similar sites) provided that care is taken to ensure that the individuals cannot be re-identified using other publicly available information.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol module indicates that 22 participants were enrolled in the study because 22 participants signed Informed Consent Documents (ICD) and screened for the study. Of the 22 participants who signed ICDs, six were excluded because they met at least one study exclusion criteria. In the Participant Flow module, we report that 16 participants Started this study because only 16 participants screened eligible and underwent training and data collection in either the control or intervention arms.
Period: Overall Study
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Started | 12 | 4
Completed | 7 | 3
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Population: To ensure consistency between the Baseline Characteristics and Outcome Measures modules in the Results Section, only the Baseline Characteristics for the 10 participants who completed the study (3 Control, 7 Powered Orthotic Exoskeleton Training Group) and whose data was analyzed (and reported in the Outcome Measures) were included in the Baseline Characteristics module of the Results Section.
Groups:
- Total: Total of all reporting groups
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 54.7 (8.4) | 62 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 3 | 10
Time Since Stroke [Mean (Standard Deviation); unit: years] | 6.6 (4.1) | 6.7 (2.1) | 6.7 (3.49)

OUTCOME MEASURES:

1. Primary Outcome: Five Times Sit to Stand Test (5xSTS)
Description: The 5xSTS is used to determine leg power and an aspect of transfer skill. This test will be used to assess a level of improved function while wearing the device. The test will also be used to assess a level of improved function not while wearing the device.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: The control group was not assessed while wearing the Powered Exoskeleton. Only the Powered Orthotic Exoskeleton Training Group was assessed while wearing the Powered Exoskeleton.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
seconds
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | -20.3 (14.2) | -10.9 (16.9)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | -9.3 (5.3) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Five Times Sit to Stand Test (5xSTS), from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.007, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.240, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Five Times Sit to Stand Test (5xSTS), from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Energy Expenditure
Description: A portable metabolic cart will assess oxygen consumption during the two ambulation conditions (i.e., with and without the device) over a 6-minute period
Time Frame: Change from Baseline after completing 36 training sessions (approximately 3 months time)
Population: Energy expenditure measurements were not conducted due to equipment malfunction of the portable metabolic cart and the inability to have it fixed during the COVID-19 pandemic. This data was not and will not be collected for this study, as the study period has concluded.
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Ratio of Stance Time of Each Limb During Ambulation
Description: Stepping parameters will be assessed using an instrumented carpet to determine if the paretic limb has more equitable and symmetrical load.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: The ratio of stance time of each limb during ambulation were not conducted due to equipment malfunction of the portable metabolic cart and the inability to have it fixed during the COVID-19 pandemic. This data was not and will not be collected for this study, as the study period has concluded
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The 6MWT was used to assess walking endurance and was conducted on a straight 12-meter length in the hospital hallway, with a small cone marking each end of the length. Participants were instructed to walk as far as possible, at a self-selected comfortable pace, for 6 minutes while a trainer followed behind them. Participants were allowed to slow down, stop, and rest if necessary if they felt fatigued during the test. The number of completed lengths (of the 12-meter stretch of the hospital hallway) was recorded and the distance in meters was calculated.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
meters
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | 59.8 (102.4) | 67 (59.4)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | 57.8 (70.4) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Six Minute Walk Test (6MWT), from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.129, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.250, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Six Minute Walk Test (6MWT), from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.073, t-test, 2 sided

5. Secondary Outcome: Ten Meter Walk Test (10MWT)
Description: The 10MWT was used to assess gait speed. Participants were instructed to walk at their own comfortable pace along a 14-meter flat course in the hospital hallway while a trainer followed behind them. The initial and final two meters were used for acceleration and deceleration, respectively, while the middle ten meters of the course were times in seconds. Participants were allowed two trails, and the fastest elapsed time was used to calculate gait speed in meters/seconds.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
meters/second
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | 0.24 (0.34) | 0.19 (0.16)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | 0.17 (0.18) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Ten Meter Walk Test (10MWT), from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.091, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.296, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Ten Meter Walk Test (10MWT), from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.427, t-test, 2 sided

6. Secondary Outcome: Timed Up and Go (TUG) Test
Description: The Timed Up and Go (TUG) Test was used as a reliable, objective measure of functional mobility. The participant was seated, with their back against the seatback, in a free-standing straight-backed chair with arms and a seat height of 17 inches. Participants were instructed to stand, walk three meters at a comfortable pace to a marked line, turn, walk back to the chair, and sit down. Timing started at the "start" command and stopped when the participant's buttocks touched the chair. Participants were allowed one practice trial prior to the timed trial.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
seconds
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | -5.9 (7.9) | -3.3 (4.9)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | -6.7 (9) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Timed Up and Go (TUG) Test, from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.063, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.447, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Timed Up and Go (TUG) Test, from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.096, t-test, 2 sided

7. Secondary Outcome: Step Length of Paretic (Pa) Lower Extremities (LE)
Description: Step lengths of the paretic (Pa) Lower Extremities were objective indices of spatiotemporal gait quality and were assessed with an instrumented pressure carpet (GaitRite Carpet, CIR Systems Inc., Franklin, NJ). Participants were instructed to walk at a comfortable, self-selected pace on a sensor equipped carpet that provided step length among other parameters. At least six consecutive steps on the carpet were needed to calculate the spatiotemporal parameters of the participant's gait.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
centimeter
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | 8.4 (15.5) | 2.2 (7.2)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | 9.3 (8) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Step Length of Paretic (Pa) Lower Extremities (LE), from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.035, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.677, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Step Length of Paretic (Pa) Lower Extremities (LE), from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.022, t-test, 2 sided

8. Secondary Outcome: Step Length of Non-paretic (NP) Lower Extremities (LE)
Description: Step lengths of the non-paretic (NP) Lower Extremities were objective indices of spatiotemporal gait quality and were assessed with an instrumented pressure carpet (GaitRite Carpet, CIR Systems Inc., Franklin, NJ). Participants were instructed to walk at a comfortable, self-selected pace on a sensor equipped carpet that provided step length among other parameters. At least six consecutive steps on the carpet were needed to calculate the spatiotemporal parameters of the participant's gait.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
centimeter
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | 6.4 (10.3) | 2.3 (2.4)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | 8.7 (5.8) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Step lengths of the non-paretic (NP) Lower Extremities (LE), from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.098, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.666, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of Step lengths of the non-paretic (NP) Lower Extremities (LE), from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.007, t-test, 2 sided

9. Secondary Outcome: Stair Climb Power Test (SCPT)
Description: The Stair Climb Power Test was used as a measure of lower extremity (LE) power and functional mobility. Participants were instructed to ascend a flight of 10 stairs as fast as possible, using the handrail as needed for safety. Participants stood at the base of the first step. Timing started on the assessor's "go" command and stopped when both feet of the participant reached the top of the tenth step.
Time Frame: Change from Baseline after completing 36 training sessions (approximately three months time)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
Number analyzed (Participants) | 7 | 3
seconds
  Change from Baseline after completing training, assessed while not wearing the Powered Exoskeleton | -7.3 (3.3) | -8.1 (5.7)
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton: number analyzed (Participants) | 7 | 0
  Change from Baseline after completing training, assessed while wearing the Powered Exoskeleton | -9.3 (7.7) |
Statistical Analysis 1: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of the Stair Climb Power Test (SCPT), from Baseline to after completing 36 training sessions. Assessed while not wearing the Powered Exoskeleton; Test type: Superiority; p = 0.001, ANOVA
Statistical Analysis 2: Comparison: Control Group; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.009, ANOVA
Statistical Analysis 3: Comparison: Powered Orthotic Exoskeleton Training Group; Within-group comparison of the Stair Climb Power Test (SCPT), from Baseline to after completing 36 training sessions. Assessed while wearing the Powered Exoskeleton; Test type: Superiority; p = 0.018, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were reported within five business days to the VA's Institutional Review Board (IRB) via an Adverse Event form and were also included on the Adverse Events log on the annual continuing review application in accordance with VA IRB policy. Adverse event data were collected through study completion, up to four months (three months of training sessions plus one month post cessation of training).
Arm/Group | Powered Orthotic Exoskeleton Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 3/12 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Powered Orthotic Exoskeleton Training Group (N=12) | Control Group (N=4)
Increased pain on the right side after using the Powered Orthotic Exoskeleton (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — After using the Keeogo device, participant stated that they had increased pain on the right side. Study physician examined the participant. Participant stated that they have this pain chronically and is associated with activity.
Cataract Procedure (Surgical and medical procedures) | 0 (0) | 1 (1) — Subject underwent two separate cataract procedures, one for each eye. Prior to requiring the procedure, the subject only completed two training sessions. As a result, the subject was placed on hold until medical clearance from the study physician.
Fall, Taken Place Outside of the Subject's Participation in Research (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — The fall took place at a restaurant when the subject was standing up from their chair. According to the participant, they had bruising on one side of the body and some minor scrapes on the other side.
Epigastric Pain and Dizziness, Taken Place Outside of the Subject's Participation in Research (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Participant had complaints of epigastric pain and dizziness since waking up. When the participant reported to a medical appointment, their provider sent them to the Emergency Department (ED). They were evaluated and left the ED in stable condition.
Fall, Taken Place During the Subject's Participation in Research (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — During study visit, the participant stumbled on the stairwell landing and caught themselves with arms and assistance from the trainer. No loss of consciousness. The participant was immediately able to right themselves and continue walking/stepping.
Loss of Consciousness due to Urinary Tract Infections (Renal and urinary disorders) | 1 (1) | 0 (0) — While at home, the subject lost consciousness for about 5 seconds. After regaining consciousness, they returned to being fully alert. They went to the emergency room and determined that the loss of consciousness was due to a urinary tract infection.

LIMITATIONS AND CAVEATS:
We were approved to begin this study during the summer of 2020, which was during the first wave of the COVID-19 pandemic. Due to the lockdown status of our VAMC at that time, no participants were permitted to be enrolled. In late April 2021, most restrictions were lifted at our VAMC, and we were able to begin the process of enrolling the targeted number of participants. The delayed start to study procedures, however, led to a smaller than anticipated number of subjects available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04241848/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04241848/ICF_000.pdf